CLINICAL TRIAL: NCT05811143
Title: Examining the Effects of Dorsal Column Stimulation on Pain From Lumbar Spinal Stenosis Related to Epidural Lipomatosis.
Status: Completed | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY20200036
Record Dates: First submitted 2023-03-20; First posted 2023-04-13 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Lipomatosis; Low Back Pain
MeSH Terms: conditions — Lipomatosis; Low Back Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Spinal Cord Stimulator — SOC Implantation of Spinal Cord Stimulator for Lipomatosis and Low Back Pain.

SUMMARY:
The specific aims of this proposal are to:

Examining the effects of dorsal column stimulation on pain from lumbar spinal stenosis related to lumbar epidural lipomatosis. The primary outcome will be improvement in VAS score of combined back and leg pain at 6 weeks follow-up. Secondary outcomes will include improvement in Visual Analog Scale (VAS) back pain scores, VAS leg pain scores, and Oswestry Disability Index (ODI) , as well as SCS complication rate.

The specific aims of this proposal are to:

Examining the effects of dorsal column stimulation on pain from lumbar spinal stenosis related to lumbar epidural lipomatosis. The primary outcome will be improvement in VAS score of combined back and leg pain at 6 weeks follow-up. Secondary outcomes will include improvement in VAS back pain scores, VAS leg pain scores, and Oswestry Disability Index, as well as SCS complication rate.

ELIGIBILITY:
Inclusion Criteria:

1. - Have chronic pain for >3 months
2. Age 18-65 years
3. Have been scheduled to be implanted with the spinal cord stimulator due to epidural lipomatosis.
4. MRI evidence of lumbar spinal stenosis with grade I-III Lumbar epidural lipomatosis and concordant history and physical examination

Exclusion Criteria:

* No evidence of lumbar epidural lipomatosis based on MRI 2. Presence of a pacemaker/ICD (to avoid possible side-effects of electrical stimulation) 3. Coagulopathy (either non-pharmacological or unable to discontinue anticoagulation due to underlying comorbidities as deemed by prescribing physician) 4. Unable to follow commands or provide consent. 5. Are not medically/psychologically stable 6. Have clinical/EMG documented motor dysfunction and have not been evaluated by spine surgeon. 7. Inappropriate surgical candidates as determined by the individual implanting physician. 8. History of laminectomy/fusion in thoracic or lumbar spine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 20 subjects who present to University Hospital Pain Medicine clinics
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
VAS-Visual Analog Scale- score of combined back and leg pain at 6 weeks follow-up. | 6 weeks
  0 meaning No Pain, 10 being worst possible pain. Higher pain means worse outcome.

SECONDARY OUTCOMES:
Change in VAS-Visual Analog Scale- score of low back pain. | 6 months, 12 months
  0 meaning No Pain, 10 being worst possible pain. Higher pain score means worse outcome.
Change in VAS-Visual Analog Scale - score of leg pain score | 6 months, 12 months
  0 meaning No Pain, 10 being worst possible pain. Higher pain score means worse outcome.
Change in Oswestry Disability Index. | 6 weeks, 6 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Salim Hayek, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals, Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No